CLINICAL TRIAL: NCT03276169
Title: Left Atrial Function Changes After Left Atrial Appendage Closure in Patients With Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xierqdoctorLAAC
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; left atrial appendage closure; left atrial function
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A total of 105 patients with persistent atrial fibrillation(AF), who are persistented more than one year and planned to undergo surgical treatment, will be allocated into two groups. These patients will receive left atrial appendage closure, radiofrequency ablation under the guidance of 3D mapping and left atrial appendage closure combined with radiofrequency ablation, respectively (allocation ratio, 1:1:1).
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will participate in the operation to record operative parameters such as LA pressure. Other researchers including follow-up personnel and the ultrasonic data analyst are uninformed about the random situation of the patients (patient information is recorded according to the random number. Random numbers corresponding to the random allocation list are stored in the research center. After follow-up of the last patient is completed, the random allocation list is published by the random number designer; and the designer does not participate in the data collection and statistics.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Left atrial appendage closure group (Experimental)
  Interventions: Procedure: Left atrial appendage closure
- Radiofrequency ablation group (Other)
  Interventions: Procedure: Radiofrequency ablation
- LAAC combined with radiofrequency ablation group (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation group

INTERVENTIONS:
Procedure: Left atrial appendage closure — Left atrial appendage closure is performed using a single endocardial plug devices guided by fluoroscopic guidance and transesophageal echocardiography
  Arms: Left atrial appendage closure group
Procedure: Radiofrequency ablation — Each patient with persistent AF receives circumferential pulmonary vein isolation under the 3D electro-anatomical mapping system , and no additional ablation is performed in the extrapulmonary sites unless the patient is diagnosed with atrial flutter before the operation.
  Arms: Radiofrequency ablation group
Procedure: LAAC combined with radiofrequency ablation group — Each patient received the same group of patients with simple radiofrequency ablation radiofrequency ablation treatment at the same time, the transcatheter occlusion of left atrial appendage opening
  Arms: LAAC combined with radiofrequency ablation group

SUMMARY:
A total of 105 patients with persistent atrial fibrillation(AF), that lasting longer than one year and planned to undergo surgical treatment, will be allocated into three groups. These patients will receive left atrial appendage closure(LAAC), radiofrequency ablation under the guidance of 3D mapping and LAAC combined with radiofrequency ablation, respectively (allocation ratio, 1:1:1). Real-time 3D ultrasound and 2D ultrasound examinations and measurement of left ventricle(LV) and left atrial(LA) function are carried out for all patients before the operation, and at 1, 2, 3 and 4 weeks and 2, 3, 6, 9 and 12 months after the operation. All ultrasound data will be stored and a professional director from the ultrasound room will be invited for quantitative analysis. Indicators for ultrasonography include: LV ejection fraction(LVEF), LV end-diastolic volume, Stroke volume, left atrial anterior and posterior diameter, left atrial volume, left atrial volume index, mitral e ", E peak, A peak, velocity time integral (VTI), left atrial ejection fraction, left atrial strain, and strain rate. Blood samples are extracted in all patients to detect type B natriuretic peptide before the operation and at 1, 2, 3 days and 1,3,6,12 months after the operation. Blood samples are extracted in all patients to detect routine blood, coagulation, D-D dimmer,Inflammatory markers (hsCRP） and other biochemical parameters before the operation and at 1, 2, 3 and 4 weeks and 1, 2, 3,6and 12 months after the operation. At the same time in operation LA pressure in all patients will be measured preoperatively and postoperatively. This study will clarify the short-term and long-term changes of LA pressure and function of patients with persistent AF after LAAC, and whether changes in left atrial pressure and function are related to inflammation indicators. This study will also to observe whether the coagulation indexes changed after LAAC that can be used to know whether the LAAC activates the coagulation system. In addition, this study to investigate the effects of radiofrequency ablation combined with LAAC on left atrial pressure and function, changes of blood coagulation and inflammatory markers, and to analyze the above findings. At an average follow-up of one year, changes in left atrial function, inflammation, coagulation, and embolic events were analyzed early (3 months after surgery) and late (1 years after surgery).

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation episode occurs in the patient that lasting longer than one year,
* atrial fibrillation cannot be prevented in patients who orally take class I and III antiarrhythmic drugs,
* and patient age is <80 years.

Exclusion Criteria:

* patients with previous history of atrial fibrillation ablation, atrial thrombosis, or valvular heart disease (moderate and severe valvular stenosis, severe valvular regurgitation),
* patients who underwent prosthetic heart valve replacement,
* pregnant women,
* patients with existing liver and kidney disease, malignant tumors or hematological system diseases.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Left atrial function of postoperative left atrial appendage occlusion detected | 1-12 month
  Transthoracic ultrasound

SECONDARY OUTCOMES:
Plasma biomarkers of inflammation assessed | 1-12 month
  Blood samples are extracted in all patients for the detection of the C reactive protein, white blood cell，red blood cell, Platelets，neutrophile and lymphocytes.
B natriuretic peptide assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Coagulation index assessed | 1-6 month
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China